CLINICAL TRIAL: NCT02426749
Title: Treatment and Recovery Monitoring of Post Traumatic Brain Injury (TBI) Symptoms
Brief Title: Treatment and Recovery Monitoring of Post TBI Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2015:032
Record Dates: First submitted 2015-04-16; First posted 2015-04-27 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2016-10

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Coil (Active Comparator): Participants of this arm will receive active rTMS intervention (treatment).
  Interventions: Device: Active repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham (Sham Comparator): Participants of this arm will receive sham rTMS intervention (treatment).
  Interventions: Device: Sham repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Active repetitive Transcranial Magnetic Stimulation (rTMS) — The treatments will be administered daily (five days/week) for two weeks, followed by three days on the third week (total of 13 treatments). Patients of both real and sham treatment groups will undergo rTMS treatment of 1.5-second duration trains of pulses at 20 Hz for a total of 25 trains with intertrain interval of 10 seconds applied to DLPFC bilaterally at 100% of the resting motor threshold. Thus, there will be a total of 1500 pulses per two sides of the brain per day, which is well within the safety limit of the rTMS application. During the intertrain intervals, the patients will be presented a series of objects and actions and asking to name them. The images will be projected on the wall in front of patient with duration of three seconds for each image. The aim is to keep the brain active while we stimulate it with rTMS.
  Arms: Active Coil
Device: Sham repetitive Transcranial Magnetic Stimulation (rTMS) — Sham rTMS is similar to Active rTMS but instead of a real coil, it uses a coil that attenuates the pulses such that no current will be induced in the brain.
  Arms: Sham

SUMMARY:
This proposal aims to investigate the effect of a promising treatment for persistent post Traumatic Brain Injury (TBI) symptoms, and to monitor TBI patient's recovery by an objective technique along with standard clinical assessments. The treatment tool is the application of repetitive Transcranial Magnetic Stimulation (rTMS) to the dorsolateral prefrontal cortex (DLPFC) of the brain. The treatment efficacy and monitoring TBI patients' recovery will be objectively assessed using Electrovestibulography (EVestGTM); this will be in parallel with clinical and standard assessments.

DETAILED DESCRIPTION:
TBI is a significant health problem mainly because of its plausible prolonged sequelae and lack of objective measures for recovery. The conventional treatment after a TBI is physical rehabilitation that helps with motor functional recovery. However, there are usually some disabling persistent post-TBI symptoms (mostly neurological) that do not respond to the current clinical and physical rehabilitation. rTMS, on the other hand, is a promising, well-tolerated, non-invasive brain neuromodulation technique that has emerged as a therapeutic tool for a variety of neurological conditions. Thus, the researchers' aim to investigate the effect of rTMS treatment on post-TBI symptoms in patients identified by the medical collaborators (Drs. Mansouri and Salter). Equally important is to have an objective measure of treatment efficacy and patient's symptoms recovery. EVestGTM is a noninvasive technique to record neural activity from the vestibular apparatus and vestibular nuclei in the external ear. After a head injury, people commonly experience balance (vestibular) problems and dizziness, as well as confused thinking. Considering the well-known bidirectional anatomical links of the vestibular system, following an impact TBI, EVestG signals are expected to change, and our pilot studies show a great potential of EVestG to monitor the impact of TBI. Thus, the researchers aim to use EVestG as an objective measure to monitor the recovery path during and after the rTMS treatment in parallel to clinical and neuro-psychological assessments.

ELIGIBILITY:
Inclusion Criteria for patients:

1. Participants must be of age 18-70 years, and have had TBI in the last 12 months prior to inclusion and presence of persistent TBI symptoms at the time of inclusion as confirmed by the co-investigator physicians.

Exclusion Criteria:

1. Use of neuro- or psycho-active medications as published in recommendations
2. Active use of illicit drugs
3. History of epilepsy
4. History of any other brain lesions including tumors, infectious, vascular, or metabolic lesions
5. Severe or recent heart diseases
6. Alcoholism
7. Pregnancy
8. The presence of metallic objects in the body; dental implants are fine but people with pacemakers are to be excluded; anything that is unsafe under MRI would be considered unsafe for TMS [26].
9. Lack of ability to adequately communicate (understand, read, speak) in English and understand the experimental protocol.
10. Pending litigation (i.e., patients with pending actions regarding disability reports, litigation, or other kinds of financial compensation).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Center, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moussavi Z, Suleiman A, Rutherford G, Ranjbar Pouya O, Dastgheib Z, Zhang W, Salter J, Wang X, Mansouri B, Lithgow B. A Pilot Randomised Double-Blind Study of the Tolerability and efficacy of repetitive Transcranial Magnetic Stimulation on Persistent Post-Concussion Syndrome. Sci Rep. 2019 Apr 2;9(1):5498. doi: 10.1038/s41598-019-41923-6. PMID 30940870

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Coil: Participants of this arm received active rTMS intervention (treatment).
  Active repetitive Transcranial Magnetic Stimulation (rTMS): The treatments were administered daily (five days/week) for two weeks, followed by three days on the third week (total of 13 treatments). Patients of both real and sham treatment groups received rTMS treatment of 1.5-second duration trains of pulses at 20 Hz for a total of 25 trains with intertrain interval of 10 seconds applied to DLPFC on the left side at 100% of the resting motor threshold. Thus, there was a total of 750 pulses per day, which was well within the safety limit of the rTMS application.
- Sham: Participants of this arm received sham rTMS intervention (treatment).
  Sham repetitive Transcranial Magnetic Stimulation (rTMS): Sham rTMS was similar to Active rTMS but instead of a real coil, it used a coil that attenuates the pulses such that no current will be induced in the brain.
Period: Overall Study
Arm/Group | Active Coil | Sham
Started | 12 | 10
Completed | 9 | 9
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Coil | Sham | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (16.1) | 53.4 (9.2) | 50.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 9 | 18
MoCA score [Mean (Standard Deviation); unit: units on a scale] — MoCA stands for Montreal Cognitive Assessment. It is a measure of cognitive ability. The scale ranges from 0 to 30, with higher scores representing better cognition.
  units on a scale | 28.1 (1.17) | 27.1 (2.98) | 27.6 (2.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in RPQ Score at Post-treatment Sessions
Description: RPQ is the Rivermead Post Concussion Symptoms Questionnaire. Scale ranges from 0 to 64 points, with higher scores representing a greater number or severity of reported symptoms.
Time Frame: Immediately following treatment (4 weeks after baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Coil | Sham
Number analyzed (Participants) | 9 | 9
units on a scale | -4.6 (10.2) | -3.4 (10.5)

2. Primary Outcome: Change From Baseline in EVestG Field Potential's Features at Post Treatment Sessions
Description: EVestG is the Electrovestibulography assessment, in which features of the neural field potential are extracted. The measurement here is a calculation of the area under the AP curve. The area is a product of the number of samples (1 / 41667 s each) and the normalized voltage (normalized so the field potential peak has a magnitude of 1). The result is summed over all detected field potentials. Due to the normalization, in a practical sense this value gives a metric of how wide or narrow the calculated field potential shape is.
Time Frame: Immediately following treatment (4 weeks after baseline)
Measure: Mean (Standard Deviation); unit: product of normalized voltage & samples
Arm/Group | Active Coil | Sham
Number analyzed (Participants) | 9 | 9
product of normalized voltage & samples | 5.64 (10.75) | 3.08 (7.01)

3. Secondary Outcome: Change From Baseline in MoCA Score at Post-treatment Sessions.
Description: MoCA is the Montreal Cognitive Assessment; the scale ranges from 0 to 30 points. Higher scores indicate a higher cognitive ability.
Time Frame: Immediately following treatment (4 weeks after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Coil | Sham
Number analyzed (Participants) | 9 | 9
score on a scale | 0.33 (1.73) | 0.67 (2.06)

4. Secondary Outcome: Change From Baseline in MADRS Score at Post-treatment Sessions
Description: MADRS is the Montgomery Asberg Depression Rating Scale. Scores range from 0 to 60, with higher scores meaning that the subject has a higher degree of depression.
Time Frame: Immediately following treatment (4 weeks after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Coil | Sham
Number analyzed (Participants) | 9 | 9
score on a scale | -3.22 (4.87) | -2.33 (7.42)
Statistical Analysis 1: Comparison: Active Coil vs Sham; Test type: Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Active Coil | Sham
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Coil (N=9) | Sham (N=9)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT02426749/Prot_SAP_000.pdf